CLINICAL TRIAL: NCT05550532
Title: A Randomized, Double-blind, Multicenter, Parallel-group, Placebo-controlled Study to Evaluate the Efficacy, Safety, and Tolerability of Aticaprant 10 mg as Adjunctive Therapy in Adult Participants With Major Depressive Disorder (MDD) With Moderate-to-severe Anhedonia and Inadequate Response to Current Antidepressant Therapy
Brief Title: A Study of Aticaprant 10 Milligrams (mg) as Adjunctive Therapy in Adult Participants With MDD With Moderate-to-severe Anhedonia and Inadequate Response to Current Antidepressant Therapy
Acronym: VENTURA-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR109230; 67953964MDD3002 (Other: Janssen Research & Development, LLC); 2022-000461-41 (EudraCT Number)
Record Dates: First submitted 2022-09-20; First posted 2022-09-22 (Actual); Results first posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Depressive Disorder, Major; Anhedonia
MeSH Terms: conditions — Depressive Disorder, Major; Anhedonia | interventions — Aticaprant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Aticaprant (Experimental): Participants will receive Aticaprant 10 milligrams (mg) tablet orally, once daily for 42 days during double-blind (DB) treatment phase in addition to their current antidepressant selective serotonin reuptake inhibitor/serotonin-norepinephrine reuptake inhibitor (SSRI/SNRI) therapy. Participants who will complete the DB treatment phase (Day 43) may be eligible to participate in a separate 52-week open-label long-term safety study 67953964MDD3003.
  Interventions: Drug: Aticaprant
- Placebo (Placebo Comparator): Participants will receive matching placebo tablet orally, once daily for 42 days during DB treatment phase in addition to their current antidepressant SSRI/SNRI therapy. Participants who will complete the DB treatment phase (Day 43) may be eligible to participate in a separate 52-week open-label long-term safety study 67953964MDD3003.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Aticaprant — Aticaprant tablet will be administered orally.
  Other Names: JNJ-67953964
  Arms: Aticaprant
Other: Placebo — Placebo tablet will be administered orally.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy of aticaprant compared with placebo as adjunctive therapy to an antidepressant in improving depressive symptoms in adult participants with major depressive disorder (MDD) with moderate to severe anhedonia (ANH+) who have had an inadequate response to current antidepressant therapy with a selective serotonin reuptake inhibitor (SSRI) or serotonin-norepinephrine reuptake inhibitor (SNRI).

DETAILED DESCRIPTION:
Depression is a common and serious psychiatric disorder which is a leading cause of disability worldwide and is associated with elevated mortality and suicide risk. Aticaprant (JNJ-67953964) is a once daily, highly selective kappa opioid receptor (KOR) antagonist, with demonstrated selectivity over mu opioid receptor (MOR) and delta opioid receptor (DOR) being developed for adjunctive treatment of MDD with ANH+. The total duration of the study will be up to 87 days. Safety evaluation including adverse events, physical examinations, urine drug test, alcohol breath tests and clinical laboratory tests will be assessed at specific time points during this study.

ELIGIBILITY:
Inclusion Criteria:

* Be medically stable on the basis of physical examination, medical history, vital signs, and 12-lead electrocardiogram (ECG) performed at screening and baseline
* Have a Hamilton depression rating Scale 17 item (HDRS-17) total score of 20 or higher at the first and second screening interviews and must not demonstrate a clinically significant improvement (that is, an improvement of more than 20 percent [%] on their HDRS-17 total score) between the first and the second independent HDRS-17 assessments
* Meet Diagnostic and Statistical Manual of Mental Disorders-5th edition (DSM-5) diagnostic criteria for recurrent or single episode major depressive disorder (MDD), without psychotic features, based upon clinical assessment and confirmed by the structural interview for DSM-5 Axis I disorders-clinical trials version (SCID-CT). Participants 65 years of age or older must have had the first onset of depression prior to 55 years of age
* Is currently receiving and tolerating well any one of the following selective serotonin reuptake inhibitor (SSRI) or serotonin-norepinephrine reuptake inhibitor (SNRI) for depressive symptoms at screening, in any approved formulation and available in the participating country/territory: citalopram, duloxetine, escitalopram, fluvoxamine, fluoxetine, milnacipran, levomilnacipran, paroxetine, sertraline, venlafaxine, desvenlafaxine at a stable dose (at or above the minimum therapeutic dose per Massachusetts General Hospital Antidepressant Treatment Response Questionnaire [MGH-ATRQ] for at least 6 weeks. The current antidepressant cannot be the first antidepressant treatment for the first lifetime episode of depression
* Participant's current major depressive episode, and antidepressant treatment response in the current depressive episode, must all be confirmed by the Site Independent Qualification Assessment

Exclusion Criteria:

* Have had in the current depressive episode, no response (treatment failure) to 5 or more antidepressant treatments including the current SSRI/SNRI (that is, the one presumed to be continued in the treatment phase) assessed using the MGH-ATRQ
* Has a history or evidence of clinically meaningful noncompliance with current antidepressant therapy
* Has a history of moderate-to-severe substance use disorder including alcohol use disorder according to diagnostic and statistical manual of mental disorders-5th edition (DSM-5) criteria within 6 months before screening
* Has had in the current episode an inadequate response to adequate course of intravenous or intranasal ketamine or esketamine, electroconvulsive therapy (that is, at least 7 treatments), vagal nerve stimulation, or deep brain stimulation device
* Has current, or a history (past 6 months), of seizures
* Has a current homicidal ideation/intent, per the investigator's clinical judgment, or has suicidal ideation with some intent to act within 3 months prior to the start of the Screening Phase, per the investigator's clinical judgment or based on the Columbia Suicide Severity Rating Scale (C-SSRS), corresponding to a response of "Yes" on Item 4 (active suicidal ideation with some intent to act, without specific plan) or Item 5 (active suicidal ideation with specific plan and intent), or a history of suicidal behavior within the past 6 months prior to the start of the Screening Phase. Participants reporting suicidal ideation with intent to act or suicidal behavior at baseline should be excluded
* Has one or more of the following diagnoses: a) A diagnostic and statistical manual of mental disorders-5th edition (DSM-5) diagnosis (which has been the primary focus of psychiatric treatment within the past 2 years) of any of the following: panic disorder, generalized anxiety disorder social anxiety disorder, specific phobia; b) A current (in the past year) DSM-5 diagnosis of: obsessive-compulsive disorder (OCD), post-traumatic stress disorder (PTSD), anorexia nervosa, bulimia nervosa; c) A current or prior (lifetime) DSM-5 diagnosis of: a psychotic disorder or major depressive disorder (MDD) with psychotic features, bipolar or related disorders, intellectual disability, autism spectrum disorder, borderline personality disorder, antisocial personality disorder, histrionic personality disorder, narcissistic personality disorders, somatoform disorders

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 444 (Actual)
Dates: Start 2022-12-06 (Actual); Primary Completion 2024-11-08 (Actual); Study Completion 2024-11-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (132):
- United States (51):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Sunwise Clinical Research, Lafayette, California
  - Pacific Neuropsychiatric Specialists, Orange, California
  - Prospective Research Innovations Inc, Rancho Cucamonga, California
  - University of California San Diego Medical Center, San Diego, California
  - CMB Clinical Trials, Santee, California
  - California Neuroscience Research, Sherman Oaks, California
  - Pacific Clinical Research Medical Group, Upland, California
  - Next Level Clinical Trials, LLC, West Covina, California
  - MCB Clinical Research Centers LLC, Colorado Springs, Colorado
  - CNS Clinical Research Group, Coral Springs, Florida
  - Sarkis Clinical Trials, Gainesville, Florida
  - New Life Medical Research Center, Inc., Hialeah, Florida
  - K2 Medical Research, Maitland, Florida
  - Vital Care Research, Miami, Florida
  - Global Medical Institutes, Miami, Florida
  - LCC Medical Research Institute Inc, Miami, Florida
  - Florida Research Center Inc., Miami, Florida
  - Ezy Medical Research, Miami, Florida
  - Felicidad Medical Research, Miami, Florida
  - Bravo Health Care Center, North Bay Village, Florida
  - APG Research LLC, Orlando, Florida
  - Combined Research Orlando, Orlando, Florida
  - Quantum Laboratories, Pompano Beach, Florida
  - CDC Research Institute LLC, Port Saint Lucie, Florida
  - Psychiatric Medicine Associates, Skokie, Illinois
  - Tandem Clinical Research, Marrero, Louisiana
  - CBH Health, Gaithersburg, Maryland
  - Michigan Clinical Research Institute, Ann Arbor, Michigan
  - Revive Research Institute, Farmington Hills, Michigan
  - Midwest Research Group, Saint Charles, Missouri
  - Premier Psychiatric Research Institute, LLC, Lincoln, Nebraska
  - Erie County Medical Center, Buffalo, New York
  - Manhattan Behavioral Medicine, New York, New York
  - New Hope Clinical Research, Charlotte, North Carolina
  - Monroe Biomedical Research, Monroe, North Carolina
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Wexner Medical Center at the Ohio State University, Columbus, Ohio
  - Conrad Clinical Research, Edmond, Oklahoma
  - Sooner Clinical Research, Oklahoma City, Oklahoma
  - Paradigm Research Professionals, LLC, Oklahoma City, Oklahoma
  - Lehigh Center for Clinical Research LLC, Allentown, Pennsylvania
  - Global Medical Institutes, Moosic, Pennsylvania
  - Clinical Trials of South Carolina, Charleston, South Carolina
  - Donald J Garcia Jr MD PA, Austin, Texas
  - Relaro Medical Trials, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - R and H Clinical Research, Stafford, Texas
  - Cedar Psychiatry, Murray, Utah
  - Northwest Clinical Research Center, Bellevue, Washington
  - Core Clinical Research, Everett, Washington
- Argentina (9):
  - Fundacion para el Estudio y Tratamiento de las Enfermedades Mentales, Buenos Aires
  - CEN Consultorios Especializados en Neurociencias, Córdoba
  - Instituto Medico DAMIC, Córdoba
  - Centro Medico Luquez, Córdoba
  - INSA Instituto de Neurociencias San Agustín, La Plata
  - Clinica Privada de Salud Mental Santa Teresa de Ávila, La Plata
  - C I A P Centro de investigacion y Asistencia en Psiquiatria, Rosario
  - Clinica Mayo de UMCB, San Miguel de Tucumán
  - Clinica El Jardin, Santiago del Estero
- Brazil (3):
  - Trial Tech Tecnologia em Pesquisas com Medicamentos, Curitiba
  - Associacao Hospitalar Moinhos de Vento, Porto Alegre
  - CEMEC - Centro Multidisciplinar de Estudos Clínicos, São Bernardo do Campo
- Bulgaria (5):
  - MHC - Sofia, EOOD, Sofia
  - DCC 'Sv. Vrach and Sv. Sv. Kuzma and Damyan', OOD, Sofia
  - Medical Center Hera EOOD, Sofia
  - Medical Center Intermedica, OOD, Sofia
  - Diagnostic Consulting Center Mladost - M Varna, Varna
- Canada (2):
  - Alpha Recherche Clinique, Québec, Quebec
  - DIEX Recherche Sherbrooke Inc, Sherbrooke, Quebec
- China (17):
  - Hebei Mental Health Center, Baoding
  - Beijing Anding Hospital of Capital Medical University, Beijing
  - Beijing Huilongguan Hospital, Beijing
  - Peking University Sixth Hospital, Beijing
  - The second Xiangya Hospital of Central South University, Changsha
  - West China Hospital Sichuan University, Chengdu
  - Guangdong Provincial People's Hospital, Guangzhou
  - Huzhou third people's Hospital, Huzhou
  - Shanghai Mental Health Center, Shanghai
  - Tongji Hospital of Tongji University, Shanghai
  - The First Hospital of Hebei Medical University, Shijiazhuang
  - Suzhou Guangji Hospital, Suzhou
  - Tianjin Anding Hospital, Tianjin
  - Wuhan Mental Health Center, Wuhan
  - Wuhu Hospital of Beijing Anding hospital, Wuhu
  - XiAn Mental Healthcare Center, Xi'an
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou
- Czechia (4):
  - Psychiatricka ambulance, MUDr. Marta Holanova, Brno
  - Neuroterapie KH S R O, Kutná Hora
  - Medical Services Prague S R O, Prague
  - Institut Neuropsychiatricke pece, Prague
- France (6):
  - CHU de Brest - Hopital de la Cavale Blanche, Bohars
  - CHU Clermont-Ferrand - Hopital Gabriel Montpied, Clermont-Ferrand
  - Cabinet Medical des Drs Prizac-Desbonnet Scottez, Douai
  - CHU de Nantes hotel Dieu, Nantes
  - Hopital Sainte Anne, Paris
  - CHRU de Tours Clinique Psychiatrique Universitaire, Tours
- Poland (4):
  - Clinsante Osrodek Badan Klinicznych, Bydgoszcz
  - Centrum Medyczne Care Clinic Katowice, Katowice
  - Filip Rybakowski Specjalistyczna Praktyka Lekarska, Poznan
  - Indywidualna Specjalistyczna Praktyka Lekarska Agnieszka Remlinger Molenda, Suchy Las
- Slovakia (8):
  - Psychomed-Svatosavsky, s.r.o., Banská Bystrica
  - Nemocnica s poliklinikou Prievidza so sidlom v Bojniciach, Bojnice
  - Psychiatricka Ambulancia Mentum S.R.O., Bratislava
  - Epamed sro, Košice
  - Univerzitna nemocnica L. Pasteura Kosice, Košice
  - Liptovska Nemocnica S Poliklinikou Mudr. Ivana Stodolu, Liptovský Mikuláš
  - Psychiatricka Ambulancia Psycholine S.R.O., Rimavská Sobota
  - Crystal Comfort s.r.o., Vranov nad Topľou
- South Africa (3):
  - Cape Town Clinical Research Centre, Cape Town
  - Gert Bosch Pretoria South Africa, Pretoria
  - Somerset West Clinical Research Unit, Strand
- South Korea (10):
  - Bucheon St. Mary's Hospital, Bucheon-si
  - Inje University Haeundae Paik Hospital, Busan
  - CHA University ilsan Medical Center, Goyang
  - Korea University Ansan Hospital, Gyeonggi-do
  - KyungHee University Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea Yeouido St. Mary's Hospital, Seoul
  - Seoul National University Hospital, Seoul
- Taiwan (4):
  - China Medical University Hospital, Taichung
  - Taipei Medical University, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Cheng Hsin General Hospital, Taipei
- United Kingdom (6):
  - University of Sussex, Brighton
  - Royal Edinburgh Hospital, Edinburgh
  - Institute of Psychiatry, London
  - Renfrewshire CMHT, Paisley
  - Moorgreen Hospital, Southampton
  - Crisis Resolution and Home Treatment Team, Wigan and Leigh

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Adult participants aged 18 to 64 years who had major depressive disorder (MDD) with or without moderate-to-severe anhedonia (ANH+ or ANH-) and elderly participants aged 65 to 74 years with MDD (ANH+ and ANH-) who had an inadequate response to an ongoing antidepressant therapy were randomized in the study.
Groups:
- Placebo: During double blind (DB) treatment phase, participants received placebo matching to aticaprant tablet orally once daily from Day 1 to Day 42 in addition to the ongoing antidepressant therapy (selective serotonin reuptake inhibitor/serotonin-norepinephrine reuptake inhibitor [SSRI/SNRI]). Participants were then followed up for safety up to 7 to 14 days after end of DB phase at Day 43 (up to Day 57). Participants who completed the DB phase (at Day 43) and were compliant to the study intervention were eligible to participate in a separate 52-week open-label long-term safety study 67953964MDD3003 (NCT05518149).
- Aticaprant 10 mg: During DB treatment phase, participants received aticaprant 10 milligrams (mg) tablet orally once daily from Day 1 to Day 42 in addition to the ongoing antidepressant therapy (SSRI/SNRI). Participants were then followed up for safety up to 7 to 14 days after end of DB phase at Day 43 (up to Day 57). Participants who completed the DB phase (at Day 43) and were compliant to the study intervention were eligible to participate in a separate 52-week open-label long-term safety study 67953964MDD3003 (NCT05518149).
Period: Overall Study
Arm/Group | Placebo | Aticaprant 10 mg
Started | 225 | 219
Participants Who Entered Follow-up Phase | 21 | 18
Completed | 211 | 209
Not Completed | 14 | 10
Not completed — Withdrawal by Subject | 8 | 3
Not completed — Adverse Event | 2 | 3
Not completed — Lost to Follow-up | 4 | 0
Not completed — Other | 0 | 4

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all randomized participants (adults and elderly) who received at least 1 dose of study intervention.
Groups:
- Placebo: During DB treatment phase, participants received placebo matching to aticaprant tablet orally once daily from Day 1 to Day 42 in addition to the ongoing antidepressant therapy (SSRI/SNRI). Participants were then followed up for safety up to 7 to 14 days after end of DB phase at Day 43 (up to Day 57). Participants who completed the DB phase (at Day 43) and were compliant to the study intervention were eligible to participate in a separate 52-week open-label long-term safety study 67953964MDD3003 (NCT05518149).
- Aticaprant 10 mg: During DB treatment phase, participants received aticaprant 10 mg tablet orally once daily from Day 1 to Day 42 in addition to the ongoing antidepressant therapy (SSRI/SNRI). Participants were then followed up for safety up to 7 to 14 days after end of DB phase at Day 43 (up to Day 57). Participants who completed the DB phase (at Day 43) and were compliant to the study intervention were eligible to participate in a separate 52-week open-label long-term safety study 67953964MDD3003 (NCT05518149).
- Total: Total of all reporting groups
Arm/Group | Placebo | Aticaprant 10 mg | Total
Number analyzed (Participants) | 223 | 217 | 440
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.3 (13.11) | 49.1 (13.14) | 49.2 (13.11)
Age, Customized [Count of Participants; unit: Participants]
  Adults (18-64 years) | 200 | 192 | 392
  From 65 to 74 years | 23 | 25 | 48
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 168 | 161 | 329
  Male | 55 | 56 | 111
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 74 | 74 | 148
  Not Hispanic or Latino | 141 | 137 | 278
  Unknown or Not Reported | 8 | 6 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 15 | 16 | 31
  Native Hawaiian or Other Pacific Islander | 2 | 1 | 3
  Black or African American | 9 | 9 | 18
  White | 182 | 177 | 359
  More than one race | 2 | 2 | 4
  Unknown or Not Reported | 13 | 11 | 24
Region of Enrollment [Count of Participants; unit: Participants]
  Argentina | 35 | 37 | 72
  Brazil | 8 | 4 | 12
  Bulgaria | 9 | 9 | 18
  Czech Republic | 11 | 7 | 18
  France | 10 | 10 | 20
  Poland | 13 | 14 | 27
  Slovakia | 19 | 17 | 36
  South Africa | 12 | 14 | 26
  Korea, Republic of | 9 | 10 | 19
  Taiwan | 3 | 2 | 5
  United Kingdom | 4 | 5 | 9
  United States | 90 | 88 | 178

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Day 43 in the Montgomery-Asberg Depression Rating Scale (MADRS) Total Score
Description: The MADRS is a clinician-rated scale designed to measure depression severity and detect changes due to antidepressant treatment. The scale consists of 10 items (apparent sadness, reported sadness, inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts, and suicidal thoughts), each of which is scored from 0 (item not present or normal) to 6 (severe or continuous presence of symptoms). MADRS total score is the sum of scores from individual question items, which ranges from 0 to 60; higher scores represent a more severe condition. Negative change in MADRS total score indicates improvement.
Time Frame: Baseline (Day 1) to Day 43
Population: Full analysis set (ANH+) included all adult randomized participants in rest of the world (ROW; countries/territories other than China) with MDD ANH+ who received at least 1 dose of study intervention. Here, 'N' (overall number of participants analyzed) signifies number of participants evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Groups:
- Aticaprant 10 mg: During DB treatment phase, participants received aticaprant 10 milligram (mg) tablet orally once daily from Day 1 to Day 42 in addition to the ongoing antidepressant therapy (SSRI/SNRI). Participants were then followed up for safety up to 7 to 14 days after end of DB phase at Day 43 (up to Day 57). Participants who completed the DB phase (at Day 43) and were compliant to the study intervention were eligible to participate in a separate 52-week open-label long-term safety study 67953964MDD3003 (NCT05518149).
Arm/Group | Placebo | Aticaprant 10 mg
Number analyzed (Participants) | 159 | 154
Units on a scale | -9.4 (0.96) | -10.0 (0.96)
Statistical Analysis 1: Comparison: Placebo vs Aticaprant 10 mg; Test type: Superiority; p = 0.670, Mixed Model for Repeated Measures Model; Least Square Mean Difference = -0.5, 95% CI 2-sided [-2.95 to 1.90], Standard Error of Mean 1.23

2. Secondary Outcome: Change From Baseline to Day 43 in Dimensional Anhedonia Rating Scale (DARS) Total Score
Description: The DARS is a 17-item self-report questionnaire that is designed to assess anhedonia in MDD across the 4 domains: hobbies, social activities, food/drink, and sensory experience. The DARS scale measures desire, motivation, effort, and consummatory pleasure. The DARS is rated on a 5-point Likert scale (0=not at all, 1=slightly, 2=moderately, 3=mostly, 4=very much) and responses are summed to generate the total score (range of 0 to 68). A lower total score is indicative of greater anhedonia. Positive changes in DARS total score indicate improvement.
Time Frame: Baseline (Day 1) to Day 43
Population: Full analysis set (ANH+) included all adult randomized participants in ROW (countries/territories other than China) with MDD ANH+ who received at least 1 dose of study intervention. Here, 'N' (overall number of participants analyzed) signifies number of participants evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Aticaprant 10 mg
Number analyzed (Participants) | 150 | 147
Units on a scale | 8.2 (1.39) | 8.8 (1.39)

3. Secondary Outcome: Change From Baseline Over Time in MADRS Total Score
Description: Change from baseline over time in MADRS total score is reported. The MADRS is a clinician-rated scale designed to measure depression severity and detect changes due to antidepressant treatment. The scale consists of 10 items (apparent sadness, reported sadness, inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts, and suicidal thoughts), each of which is scored from 0 (item not present or normal) to 6 (severe or continuous presence of symptoms). MADRS total score is the sum of scores from individual question items, which ranges from 0 to 60; higher scores represent a more severe condition. Negative change in MADRS total score indicates improvement.
Time Frame: Baseline (Day 1), Day 15, Day 29, and Day 43
Population: Full analysis set (ANH+) included all adult randomized participants in ROW (countries/territories other than China) with MDD ANH+ who received at least 1 dose of study intervention. Here, 'N' (overall number of participants analyzed) signifies participants evaluable for this outcome measure and 'n' (number analyzed) signifies number of participants analyzed at specified timepoints.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Aticaprant 10 mg
Number analyzed (Participants) | 161 | 160
Units on a scale
  Day 15 | -4.4 (0.75) | -5.4 (0.74)
  Day 29: number analyzed (Participants) | 159 | 157
  Day 29 | -7.5 (0.89) | -8.0 (0.89)
  Day 43: number analyzed (Participants) | 159 | 154
  Day 43 | -9.4 (0.96) | -10.0 (0.96)

4. Secondary Outcome: Percentage of Participants Who Achieved Response on Depressive Symptoms Scale Based on MADRS Total Score at Day 43
Description: Percentage of participants who achieved response on depressive symptoms scale based on MADRS total score at Day 43 are reported. Responders are defined as participants with a >=50 percent (%) improvement in the MADRS total score from baseline to a given timepoint. The MADRS is a clinician-rated scale designed to measure depression severity and detect changes due to antidepressant treatment. The scale consists of 10 items (apparent sadness, reported sadness, inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts, and suicidal thoughts), each of which is scored from 0 (item not present or normal) to 6 (severe or continuous presence of symptoms). MADRS total score is the sum of scores from individual question items, which ranges from 0 to 60; higher scores represent a more severe condition. Negative change in MADRS total score indicates improvement.
Time Frame: At Day 43
Population: Full analysis set (ANH+) included all adult randomized participants in ROW (countries/territories other than China) with MDD ANH+ who received at least 1 dose of study intervention.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Aticaprant 10 mg
Number analyzed (Participants) | 166 | 165
Percentage of participants | 28.3 | 27.9

5. Secondary Outcome: Percentage of Participants With Remission of Depressive Symptoms Based on MADRS Total Score at Day 43
Description: Percentage of participants with remission of depressive symptoms based on MADRS total score at Day 43 is reported. Participant is defined as a remitter at a given time point if the MADRS total score is less than or equal to (<=)10 at that time point. The MADRS is a clinician-rated scale designed to measure depression severity and detect changes due to antidepressant treatment. The scale consists of 10 items (apparent sadness, reported sadness, inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts, and suicidal thoughts), each of which is scored from 0 (item not present or normal) to 6 (severe or continuous presence of symptoms). MADRS total score is the sum of scores from individual question items, which ranges from 0 to 60; higher scores represent a more severe condition. Negative change in MADRS total score indicates improvement.
Time Frame: At Day 43
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Aticaprant 10 mg
Number analyzed (Participants) | 166 | 165
Percentage of participants | 16.3 | 15.8

6. Secondary Outcome: Change From Baseline to Day 43 in Patient Health Questionnaire, 9-Item (PHQ-9) Total Score
Description: Change from baseline to Day 43 in PHQ-9 total score is reported. The PHQ-9 is a 9-item, participant reported outcome measure to assess depressive symptoms. The scale scores each of the 9 symptom domains of the Diagnostic and Statistical Manual of Mental Disorders-5th Edition (DSM-5) MDD criteria. Each item is rated on a 4 point scale (0=not at all, 1=several days, 2=more than half the days, and 3=nearly every day). The participant's item responses are summed to provide a total score (range of 0 to 27), with higher scores indicating greater severity of depressive symptoms. The severity of the PHQ-9 is categorized as follows: none-minimal (0-4), mild (5-9), moderate (10-14), moderately severe (15-19) and severe (20-27). Negative changes in PHQ-9 total score indicate improvement.
Time Frame: Baseline (Day 1) to Day 43
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Aticaprant 10 mg
Number analyzed (Participants) | 150 | 150
Units on a scale | -5.5 (0.58) | -5.2 (0.58)
Statistical Analysis 1: Comparison: Placebo vs Aticaprant 10 mg; Test type: Superiority; Least Square Mean Difference = 0.3, 95% CI 2-sided [-1.13 to 1.71], Standard Error of Mean 0.72

7. Secondary Outcome: Change From Baseline Over Time in DARS Total Score
Description: Change from baseline over time in DARS total score is reported. The DARS is a 17-item self-report questionnaire that is designed to assess anhedonia in MDD across the 4 domains: hobbies, social activities, food/drink, and sensory experience. The DARS scale measures desire, motivation, effort, and consummatory pleasure. The DARS is rated on a 5-point Likert scale (0=not at all, 1=slightly, 2=moderately, 3=mostly, 4=very much) and responses are summed to generate the total score (range of 0 to 68). A lower total score is indicative of greater anhedonia. Positive changes in DARS total score indicate improvement.
Time Frame: Baseline (Day 1), Days 15, 29, and 43
Population: Full analysis set (ANH+) included all adult randomized participants in ROW (countries/territories other than China) with MDD ANH+ who received at least 1 dose of study intervention. Here, 'N' (overall number of participants analyzed) signifies participants evaluable for this outcome measure and 'n' (number analyzed) signifies number of participants who were analyzed at specified timepoints.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Aticaprant 10 mg
Number analyzed (Participants) | 152 | 149
Units on a scale
  Day 15 | 3.5 (1.17) | 4.2 (1.17)
  Day 29: number analyzed (Participants) | 148 | 146
  Day 29 | 6.9 (1.27) | 7.1 (1.27)
  Day 43: number analyzed (Participants) | 150 | 147
  Day 43 | 8.2 (1.39) | 8.8 (1.39)

8. Secondary Outcome: Change From Baseline Over Time in the PHQ-9 Anhedonia-specific Item (PHQ-9, Item 1)
Description: Change from baseline over time in the PHQ-9 anhedonia-specific item (PHQ-9, item 1 is little interest or pleasure in doing things) is reported. The PHQ-9 is a 9-item, participant reported outcome measure to assess depressive symptoms. The scale scores each of the 9 symptom domains of the Diagnostic and Statistical Manual of Mental Disorders-5th Edition (DSM-5) MDD criteria. Each item is rated on a 4 point scale (0=not at all, 1=several days, 2=more than half the days, and 3=nearly every day). The participant's item responses are summed to provide a total score (range of 0 to 27), with higher scores indicating greater severity of depressive symptoms. The severity of the PHQ-9 is categorized as follows: none-minimal (0-4), mild (5-9), moderate (10-14), moderately severe (15-19) and severe (20-27). PHQ-9, item 1 score ranged from 0-3. Higher score indicates more severe disease. Negative change in PHQ-9, item 1 score indicates improvement.
Time Frame: Baseline (Day 1), Day 15, Day 29, and Day 43
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Aticaprant 10 mg
Number analyzed (Participants) | 157 | 152
Units on a scale
  Day 15 | -0.4 (0.93) | -0.6 (1.08)
  Day 29: number analyzed (Participants) | 149 | 149
  Day 29 | -0.7 (1.00) | -0.8 (1.05)
  Day 43: number analyzed (Participants) | 150 | 150
  Day 43 | -0.9 (1.12) | -0.9 (1.08)

9. Secondary Outcome: Percentage of Participants With a Score Less Than (<) 2 in the PHQ-9 Anhedonia-specific Item (PHQ-9, Item 1) at Day 43
Description: Percentage of participants with a score <2 in the PHQ-9 anhedonia-specific item (PHQ-9, item 1 is little interest or pleasure in doing things) at Day 43 is reported. The PHQ-9 is a 9-item, participant reported outcome measure to assess depressive symptoms. The scale scores each of the 9 symptom domains of the Diagnostic and Statistical Manual of Mental Disorders-5th Edition (DSM-5) MDD criteria. Each item is rated on a 4 point scale (0=not at all, 1=several days, 2=more than half the days, and 3=nearly every day). The participant's item responses are summed to provide a total score (range of 0 to 27), with higher scores indicating greater severity of depressive symptoms. The severity of the PHQ-9 is categorized as follows: none-minimal (0-4), mild (5-9), moderate (10-14), moderately severe (15-19) and severe (20-27).
Time Frame: At Day 43
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Aticaprant 10 mg
Number analyzed (Participants) | 132 | 136
Percentage of participants | 50.8 | 46.3

10. Secondary Outcome: Change From Baseline Over Time in Patient Reported Outcomes Measurement Information System Short Form - Ability to Participate in Social Roles and Activities - 8a (PROMIS-APS 8a)
Description: Change from baseline over time in the PROMIS-APS 8a is reported. This 8-item measure assesses participants' ability to participate in social roles and activities. The items measures the degree of involvement in social roles, activities, and responsibilities, including work, family, friends, and leisure. Each item is rated on a 5-point ordinal scale including 1=always, 2=usually, 3=sometimes, 4=rarely and 5=never, with higher scores indicating better social functioning. The total scores of PROMIS-APS 8a are scaled on a T-score metric with a mean of 50 and a standard deviation of 10. PROMIS-APS 8a total score ranges from 8 to 40 and T-score ranges from 25.9 to 65.4, a higher score indicates better social functioning. Positive change in score indicates improvement.
Time Frame: Baseline (Day 1), Days 15, 29, and 43
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: T-score
Arm/Group | Placebo | Aticaprant 10 mg
Number analyzed (Participants) | 142 | 134
T-score
  Day 15: number analyzed (Participants) | 141 | 132
  Day 15 | 1.4 (0.54) | 1.5 (0.55)
  Day 29: number analyzed (Participants) | 139 | 130
  Day 29 | 3.2 (0.57) | 3.1 (0.59)
  Day 43 | 3.9 (0.63) | 4.3 (0.64)

11. Secondary Outcome: DB Treatment Phase: Percentage of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: Percentage of participants with TEAEs during DB treatment phase are reported. An AE is any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the intervention. TEAE is defined as any AE occurring at or after the initial administration of study intervention through the end of DB phase.
Time Frame: From start of treatment (Day 1) up to Day 43
Population: Safety analysis set included all randomized participants (adults and elderly) in ROW (countries/territories other than China) who received at least 1 dose of study intervention.
Measure: Number; unit: Percentage of participants
Groups:
- DB: Placebo: During DB treatment phase, participants received placebo matching to aticaprant tablet orally once daily from Day 1 to Day 42 in addition to the ongoing antidepressant therapy (SSRI/SNRI).
- DB: Aticaprant 10 mg: During the DB treatment phase, participants received aticaprant 10 mg tablet orally once daily from Day 1 to Day 42 in addition to the ongoing antidepressant therapy (SSRI/SNRI).
Arm/Group | DB: Placebo | DB: Aticaprant 10 mg
Number analyzed (Participants) | 223 | 217
Percentage of participants | 38.1 | 44.2

12. Secondary Outcome: Follow-up (FU) Phase: Percentage of Participants With AEs
Description: Percentage of participants with AEs during FU phase are reported. An AE is any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the intervention.
Time Frame: From Day 44 up to Day 57
Population: Follow-up analysis set included all randomized participants in ROW (countries/territories other than China) who entered the follow-up phase after the double-blind treatment phase.
Measure: Number; unit: Percentage of participants
Groups:
- FU: Placebo: Participants who received placebo and completed DB phase entered the follow-up phase and were then followed up for safety up to 7 to 14 days after end of DB phase at Day 43 (up to Day 57).
- FU: Aticaprant 10 mg: Participants who received aticaprant 10 mg and completed DB phase entered the follow-up phase and were then followed up for safety up to 7 to 14 days after end of DB phase at Day 43 (up to Day 57).
Arm/Group | FU: Placebo | FU: Aticaprant 10 mg
Number analyzed (Participants) | 21 | 18
Percentage of participants | 0 | 5.6

ADVERSE EVENTS:
Time Frame: All cause mortality: DB treatment phase: From screening (-30 days) up to Day 43, FU Phase: From Day 44 up to Day 57; Serious and Other AEs: DB phase: From Day 1 up to Day 43; FU phase: From Day 44 up to Day 57
Description: All cause mortality: All participants randomized into the study. Serious and Other AEs: DB phase: Safety analysis set included all randomized participants (adults and elderly) in ROW (countries/territories other than China) who received at least 1 dose of study treatment. FU phase population included all randomized participants in ROW (countries/territories other than China) who entered the FU phase after the double-blind treatment phase.
Groups:
- FU: Placebo: Participants who received placebo and completed DB phase entered follow-up phase and were then followed up for safety up to 7 to 14 days after end of DB phase at Day 43 (up to Day 57).
- FU: Aticaprant 10 mg: Participants who received aticaprant 10 mg and completed DB phase entered follow-up phase and were then followed up for safety up to 7 to 14 days after end of DB phase at Day 43 (up to Day 57).
Arm/Group | DB: Placebo | DB: Aticaprant 10 mg | FU: Placebo | FU: Aticaprant 10 mg
All-Cause Mortality (participants affected / at risk) | 0/225 | 0/219 | 0/21 | 0/18
Serious Adverse Events (participants affected / at risk) | 1/223 | 0/217 | 0/21 | 0/18
Other Adverse Events (participants affected / at risk) | 18/223 | 39/217 | 0/21 | 1/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DB: Placebo (N=223) | DB: Aticaprant 10 mg (N=217) | FU: Placebo (N=21) | FU: Aticaprant 10 mg (N=18)
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DB: Placebo (N=223) | DB: Aticaprant 10 mg (N=217) | FU: Placebo (N=21) | FU: Aticaprant 10 mg (N=18)
Diarrhoea (Gastrointestinal disorders) | 9 | 17 | 0 | 0
Suicidal Ideation (Psychiatric disorders) | 1 | 1 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 9 | 25 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2023-02-22): https://cdn.clinicaltrials.gov/large-docs/32/NCT05550532/Prot_000.pdf
  • Statistical Analysis Plan (2024-10-03): https://cdn.clinicaltrials.gov/large-docs/32/NCT05550532/SAP_001.pdf